CLINICAL TRIAL: NCT02037737
Title: Impact and Use of Abatacept IV for Rheumatoid Arthritis in Real Life Setting in Patients With Inadequate Response to One or Several Conventional DMARDs Including Methotrexate in France. A Database Analysis Based on the ACTION Study
Brief Title: Impact and Use of Abatacept IV for Rheumatoid Arthritis in Real Life Setting
Acronym: ReACTION
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-409
Record Dates: First submitted 2013-11-21; First posted 2014-01-16 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients on Abatacept IV: Rheumatoid Arthritis (RA) patients with inadequate response to one or more conventional DMARDs including Methotrexate and treated with Abatacept IV according to routine clinical practice in France
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept

SUMMARY:
The purpose of this study is to assess Abatacept Intravenous (IV) effectiveness in patients with inadequate response to one or more conventional Disease Modifying Against Rheumatism (DMARDs) including Methotrexate in France, through the estimation of Abatacept retention rate over 2 years and reasons of discontinuation

DETAILED DESCRIPTION:
Observational Model:

Other: ReACTION is a study using secondary data originally collected in ACTION study. In ACTION, data were collected prospectively from October 2010 up to 2015 at each clinical visit. In France, data collection started in June 2011

ELIGIBILITY:
Inclusion Criteria:

- All patients enrolled in ACTION with inadequate response to one or more conventional DMARDs including Methotrexate and treated with Abatacept IV will be included in ReACTION

ACTION inclusion criteria for France were:

* Male or female subjects of more than 18 years old
* Patients with a diagnosis of established moderate to severe active RA
* Patients who at their physician's discretion are treated with Abatacept (initiated or already on treatment within 3 months) according to routine clinical practice
* Patients for whom baseline characteristics are available
* Patients consent for usage of their data in ACTION study
* Patients who were not included in any interventional clinical trial in RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients with inadequate response to one or more conventional DMARDs including Methotrexate and treated with Abatacept IV according to routine clinical practice in France
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Abatacept IV effectiveness in patients with inadequate response to one or more conventional DMARDs including Methotrexate in France, through the estimation of Abatacept retention rate over 2 years and reasons of discontinuation | Up to 2 years of followup

SECONDARY OUTCOMES:
Abatacept effectiveness in the treated population | 3, 6, and 12 months and every 3 months up to 2 years of followup
  Based on simplified disease activity score - 28 joints (DAS28), clinical disease activity index (CDAI), health assessment questionnaire (HAQ), and occurrence of serious adverse events
Impact of patient and disease characteristics on treatment outcomes | Every 3 months up to 2 years of followup
Joint population of French patients with inadequate response to one or more conventional DMARDs including Methotrexate treated with Abatacept IV (demographics, medical history, disease characteristics, previous treatments) | Every 3 months up to 2 years of followup
Conditions of Abatacept IV utilization in first line of biologic agents (indication, dosage, administration schedule, treatment duration, concomitant treatments) | Every 3 months up to 2 years of followup
Therapeutic strategies over time including change in concomitants treatments | Every 3 months up to 2 years of followup
The healthcare resource use as assessed by number of visits to any rheumatologists, hospitalizations | Every 3 months up to 2 years of followup
Abatacept effectiveness in patients with inadequate response to one or more conventional DMARDs including Methotrexate of the patients treated with Abatacept IV according to Summary Product Characteristics (SmPC) | Every 3 months up to 2 years of followup

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb